CLINICAL TRIAL: NCT00500604
Title: A Comparative Study of the Efficacy of Irbesartan/Hydrochlorothiazide 300/25 mg Versus Valsartan/Hydrochlorothiazide 160/25 mg Using Home Blood Pressure Monitoring in the Treatment of Mild to Moderate Hypertension
Brief Title: Efficacy of Irbesartan/Hydrochlorothiazide Versus Valsartan/Hydrochlorothiazide in Mild to Moderate Hypertension
Acronym: COSIMA2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBEH_R_02584
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Hydrochlorothiazide; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): * period 1: Hydrochlorothiazide 12.5 mg for 3-5 weeks
  * period 2: One 150/12.5mg tablet every morning for 8 weeks.
  * period 3: One 300/12.5mg tablet every morning for 8 weeks.
  * period 4: Two 150/12.5mg tablets every morning for 8 weeks.
  Interventions: Drug: Irbesartan/hydrochlorothiazide; Drug: Hydrochlorothiazide
- B (Active Comparator): * period 1: Hydrochlorothiazide 12.5 mg for 3-5 weeks
  * period 2: One 80/12.5mg tablet every morning for 8 weeks.
  * period 3: One 160/12.5mg tablet every morning for 8 weeks.
  * period 4: Two 80/12.5mg tablets every morning for 8 weeks.
  Interventions: Drug: Valsartan/hydrochlorothiazide; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Irbesartan/hydrochlorothiazide — 150/12.5mg tablet and 300/12.5mg tablet
  Arms: A
Drug: Valsartan/hydrochlorothiazide — 80/12.5mg tablet and 160/12.5mg tablet
  Arms: B
Drug: Hydrochlorothiazide — 12.5 mg administered orally, once daily in the morning

SUMMARY:
The primary objective is to compare the efficacy of irbesartan/hydrochlorothiazide 300/25mg against valsartan/hydrochlorothiazide 160/25mg in reducing mean systolic blood pressure (SBP) as measured by home blood pressure monitoring (HBPM) after 24 weeks compared with baseline.

The secondary objectives are:

* To compare the percentage of patients with normal blood pressure as measured by HBPM and at the doctor's office at weeks 16 and 24
* To compare the differences in mean Diastolic Blood Pressure (DBP), mean morning and evening SBP and DBP evaluated by HBPM at weeks 16 and 24
* To compare the difference in mean SBP evaluated by HBPM at week 16
* To compare the differences in mean SBP and DBP evaluated at the doctor's office at weeks 16 and 24
* To determine the incidence and severity of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Established essential hypertension, untreated or treated but uncontrolled with treatment:

  * Office SBP ≥ 160 mmHg for untreated patients
  * Office SBP ≥ 140 mmHg for patients already treated with an antihypertensive drug.
* Previous antihypertensive therapy must have been implemented for a minimum of 4 weeks and must be either monotherapy or one of the following permitted combination drugs:

  * ACE inhibitor / calcium channel blocker
  * Beta blocker / calcium channel blocker
  * Beta blocker / low dose diuretic
  * ACE inhibitor / low dose diuretic

Exclusion Criteria:

* SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg evaluated at doctor's office at Visit 1
* Known or suspected causes of secondary hypertension
* Patient with bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, a renal transplant or only has one functioning kidney
* Type 1 diabetes mellitus
* Significant cardiovascular, neurological, endocrine, renal, metabolic, or gastrointestinal disease, a malignancy or any other diseases considered by the Investigator to make participation in the study not in the best interest of the subject
* Known hypersensitivity to diuretics or sulphonamides or history of angioedema or cough related to the administration of an angiotensin II receptor antagonist or any combination of the drugs used
* Known contraindications to any of the study drugs
* Concomitant use of any other antihypertensive treatment
* Use of any of the investigational products for this study within the 3 months prior to the study
* Inability to obtain a valid HBPM recording i.e., obesity, arm circumference > 32 cm or arrhythmia
* Administration of any other investigational drug in the last 30 days before enrolment and during the course of the study
* Pregnant or breast-feeding women
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1617 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Reduction in mean SBP as measured by HBPM | From week 0 to week 24

SECONDARY OUTCOMES:
Reduction in mean DBP as measured by HBPM | From week 0 to weeks 16 and 24
Reduction in mean morning and evening SBP as measured by HBPM | From week 0 to weeks 16 and 24
Reduction in mean morning and evening DBP as measured by HBPM | From week 0 to weeks 16 and 24
Reduction in mean SBP and mean DBP evaluated at the doctor's office | From week 0 to weeks 16 and 24
Number of normalised patients as measured by HBPM | From week 0 to weeks 16 and 24
Number of normalised patients evaluated at the doctor's office | From week 0 to weeks 16 and 24
Reduction in mean SBP as measured by HBPM | From week 0 to week 16
Adverse events, vital signs, laboratory tests | From visit 1 to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Blayney, Study Director — Sanofi
Locations (14):
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Jakarta, Indonesia
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Karachi, Pakistan
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Ho Chi Minh City, Vietnam